CLINICAL TRIAL: NCT06136325
Title: Treatment of Anal Fistulas With Obsidian RFT® - a Retrospective Analysis
Brief Title: Treatment of Anal Fistulas With Obsidian RFT®
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christopher Dawoud, Principal Investigator; MD, Medical University of Vienna
Other Study IDs: 56
Record Dates: First submitted 2023-10-29; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Anal Fistula; Minimal Invasive Surgery; Platelet-rich Fibrin Foam
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Obsidian RFP anal fistula surgery — Anal fistula closure with instillation in the fistula tract and the inner ostium of Obsidian RTF®

SUMMARY:
The study conducted a retrospective analysis from January 2018 to December 2022 on patients who received anal fistula closure with Obsidian RTF® at the Department of General Surgery, Medical University of Vienna.

DETAILED DESCRIPTION:
Anal fistulas present a significant challenge in colorectal surgery, featuring abnormal passages between the anal canal and surrounding tissues. Traditional treatments, while effective, may risk damaging the anal sphincter complex and subsequent fecal incontinence. Sphincter-preserving techniques like autologous compound platelet-rich fibrin foam have gained popularity, offering potential for better functional outcomes in anal fistula treatment. In this context, our retrospective study aims to evaluate the efficacy and safety of autologous compound platelet-rich fibrin foam, specifically Obsidian RFT®, analyzing its success in fistula closure and functional outcomes, thus contributing to the advancement of sphincter-preserving methods in anal fistula management.

The study conducted a retrospective analysis from January 2018 to December 2022 on patients who received anal fistula closure with Obsidian RTF® at the Department of General Surgery, Medical University of Vienna.

Clinical diagnosis, complemented by radiographic imaging, was employed to confirm inconclusive cases.

Demographic, comorbidity, fistula characteristics, and postoperative data were collected from electronic records.

ELIGIBILITY:
Inclusion Criteria:

* patients who received anal fistula closure with Obsidian RTF® at the Department of General Surgery, Medical University of Vienna

Exclusion Criteria:

* unclear documentation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, receiving an anal fistula closure with Obsidian RTF®, were included into the final analysis.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Closure rate anal fistula | 24 months
  anal fistula closure rate according to documentation in the patient administration system

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dawoud, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dawoud C, Girgis K, Stift A, Harpain F, Riss S. Treatment of anal fistulas with Obsidian RFT(R): just another autologous compound platelet-rich fibrin foam? Tech Coloproctol. 2024 Aug 2;28(1):93. doi: 10.1007/s10151-024-02968-6. PMID 39095560